CLINICAL TRIAL: NCT03935516
Title: Comparing Outcomes of Extended Elbow Versus Flexed Elbow Casting for Treatment of Displaced Pediatric Both Bone Forearm Fractures: A Randomized, Controlled Trial
Brief Title: Extended vs Flexed Elbow Casting
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study team had difficulties recruiting and enrolling patients into this study.
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-1056; SMPH\ORTHOPEDIC&REHAB\ORTHO (Other: UW Madison); A536110 (Other: UW Madison)
Record Dates: First submitted 2018-05-29; First posted 2019-05-02 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Fracture;Elbow
Keywords: cast; open growth plate; pediatric; both bone
MeSH Terms: conditions — Elbow Fractures | interventions — POLR1G protein, human

STUDY DESIGN:
Intervention Model Description: The study design is a prospective, randomized controlled trial comparing extended elbow and flexed elbow casting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flexed Elbow (Experimental): The first group will be placed in a cast with the elbow bent.
  Interventions: Other: Cast
- Extended Elbow (Experimental): The second will be placed in a cast with the elbow straight.
  Interventions: Other: Cast

INTERVENTIONS:
Other: Cast — The use of plaster and/or fiberglass for casting of subject arm.

SUMMARY:
The study design is a prospective, randomized controlled trial comparing extended elbow and flexed elbow casting. This study design will provide the highest quality evidence to investigate our primary hypothesis that extended elbow casting for proximal both bone forearm fractures will result in less loss of fracture alignment. The study population eligible for screening will be patients with open growth plates and both bone forearm fractures.

DETAILED DESCRIPTION:
Guardians of patients will be approached for informed consent as soon as is feasible following determination of eligibility. Injury characteristics will be obtained from the enrolling physician and the participant's medical record.

Participants will be prospectively followed at 2, 4, 6, and 24 weeks post casting. All follow-ups will occur in person in clinic and will consist of radiographs, a clinical examination and a brief interview. The follow up time points and radiographs are all part of standard clinical care. The 24 week follow up visit is an optional clinical care visit.

Study duration: 48 months; 40 month enrollment period, 6 month patient follow up and 2 month data analysis period

Sample size: 88 patients will be consented per arm.

Questionnaires: All questionnaires will take approximately 10 minutes total of the family's time. And all questionnaires for done solely for research purposes.

Treatment Crossover Cross over from one treatment arm to another should be rare. Cross over should only occur because of poor cast tolerance or inability to maintain reduction in one position vs. another. If the extension cast is unsatisfactory to the caregivers/guardians or patients they may be converted to a flexed elbow cast. These study participants will remain in the study and be included in an intention-to-treat manner in the final analysis.

To streamline the ease of randomization in a busy department like the ED, patients with an even medical record number will be enrolled in the extended elbow cast and all odd medical record number patients will be enrolled in the flexed elbow cast. All CRFs will be pre-labeled with a study ID. The research staff will then record the study ID on the paper log that is locked in the ED cabinet. The consents/assents and the eligibility checklist will be stored in a separate folder in the ED cabinet and picked up weekly by the study coordinator who will then store the consents/assents and eligibility checklist of enrolled patients in a locked filing cabinet in their Dept. of Ortho office.

All study visits coincide with regular clinic follow up. The 5 month visits is an optional clinic visit. The Demographic questionnaire (CRF 001) will be given to them at the first clinic visit. The family will be asked verbally for responses to CRF 003 regarding cast and patient experience at every clinic visit. The rest of the CRFs will be completed by study staff regarding condition of cast (CRF003), CRF002 deals with the alignment of both forearm bones via the radiograph, and CRF004 is the elbow motion evaluation done by the study staff. CRF004 is a formal measurement using a goniometer (protractor), whereas the clinical standard of care is visual assessment without the goniometer.

ELIGIBILITY:
Inclusion Criteria:

1. Both bone forearm fractures in which the fracture of the radius and/or ulna is located in the proximal one half of the bone
2. The fracture requires a reduction maneuver
3. All skeletally immature individuals under the age of 18
4. Patient aged greater than three years old
5. Patient or patient's consenting parent/guardian competent in English.

Exclusion Criteria:

1. Skeletally mature individuals
2. Both fractures are located in the distal one-half of the radius and ulna
3. Isolated fractures of the radius or ulna
4. The fracture does not require a reduction maneuver
5. Any nerve or arterial injury in the injured extremity
6. Humerus fracture on the ipsilateral side
7. Any open fracture requiring formal surgical debridement
8. Patient or patient's consenting parent/guardian not competent in English.
9. Patient or patient's consenting parent/guardian not present.

9. Severe problems with maintaining follow-up (e.g live in different state) 10. Contractures in which applying an extended elbow cast is not possible or practical

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Alignment | 6 weeks
  To compare the proportion of proximal both bone forearm fractures that have lost alignment within 6 weeks in patients treated in a flexed elbow cast compared to those treated in an extended elbow cast.

SECONDARY OUTCOMES:
Complication Rate | approximately 24 weeks
  To compare cast complication rate between those treated in cast with elbow in flexion compared to those treated with elbow in extension.
Range of Motion | 6 weeks and 24 weeks
  To compare elbow range of motion at 6 weeks and 24 weeks post-treatment between patients treated in cast with elbow in flexion compared to those treated with elbow in extension
Caregiver Satisfaction Scores | 6 weeks
  Overall condition and satisfaction of patient's cast.
  Measured by: excellent, good, average, below average, or poor.

CONTACTS AND LOCATIONS:
Locations (1):
- American Family Children's Hospital, Madison, Wisconsin, United States